CLINICAL TRIAL: NCT00133952
Title: The Effect of Ruboxistaurin on Vision Loss in Patients With Diabetes Mellitus and Clinically Significant Macular Edema
Brief Title: Effect of Ruboxistaurin on Clinically Significant Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5882; B7A-MC-MBCU (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — ruboxistaurin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Ruboxistaurin (Experimental): 32 mg taken orally daily for up to 48 months
  Interventions: Drug: Ruboxistaurin
- Placebo (Placebo Comparator): Taken orally daily for up to 48 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ruboxistaurin — Administered orally
  Other Names: LY333531
  Arms: Ruboxistaurin
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of the study is to test the hypothesis that oral administration of ruboxistaurin will reduce the occurrence of sustained moderate visual loss (SMVL) in patients with clinically significant macular edema. SMVL is defined as a 15 letter or more decrease from baseline in best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity that is sustained for the patient's last 6 months of study participation. The SMVL data from this study will be combined with the SMVL data from Study B7A-MC-MBDL for the purpose of comparing ruboxistaurin to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes
* 18 years or older
* Hemoglobin A1c (HbA1c) less than or equal to 11%
* Mild to very severe non-proliferative diabetic retinopathy in the study eye
* Clinically significant macular edema in the study eye not within 100 microns of center of macula

Exclusion Criteria:

* Previous surgery or laser treatment (or need for laser treatment within 3 months) in the study eye
* Glaucoma in the study eye
* Unstable cardiovascular disease
* Major surgery within past 3 months
* Significantly impaired kidney or liver function, or malignancy requiring chemotherapy or radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2005-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Beutner, Study Director — Chromaderm, Inc.
Locations (41):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Artesia, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portsmouth, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slingerlands, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Mifflin, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mississauga, Ontario
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glostrup Municipality
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas, Lithuania
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
- Portugal (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest, Romania
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valladolid
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Derived] Sheetz MJ, Aiello LP, Davis MD, Danis R, Bek T, Cunha-Vaz J, Shahri N, Berg PH; MBDL and MBCU Study Groups. The effect of the oral PKC beta inhibitor ruboxistaurin on vision loss in two phase 3 studies. Invest Ophthalmol Vis Sci. 2013 Mar 11;54(3):1750-7. doi: 10.1167/iovs.12-11055. PMID 23404115
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ruboxistaurin: 32 milligrams (mg) taken orally daily for up to 48 months
Period: Overall Study
Arm/Group | Placebo | Ruboxistaurin
Started | 157 | 152
Received at Least One Dose of Study Drug | 153 | 149
Completed | 115 | 124
Not Completed | 42 | 28
Not completed — Adverse Event | 1 | 2
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 9 | 14
Not completed — Protocol Entry Criteria Exclusion | 4 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 20 | 4
Not completed — Physician Decision | 4 | 3
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ruboxistaurin | Total
Number analyzed (Participants) | 157 | 152 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.3) | 55.4 (9.9) | 55.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 133
  Male | 90 | 86 | 176
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 117 | 111 | 228
  African Descent | 18 | 15 | 33
  East Asian | 2 | 3 | 5
  West Asian | 0 | 2 | 2
  Hispanic | 20 | 21 | 41
Region of Enrollment [Number; unit: participants]
  United States | 52 | 46 | 98
  Portugal | 16 | 17 | 33
  Mexico | 7 | 10 | 17
  Canada | 11 | 11 | 22
  Spain | 9 | 9 | 18
  Lithuania | 1 | 0 | 1
  Romania | 13 | 12 | 25
  Denmark | 26 | 26 | 52
  Germany | 13 | 10 | 23
  United Kingdom | 5 | 5 | 10
  France | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Moderate Visual Loss (SMVL) Any Time Baseline Through Month 48
Description: SMVL is defined as a 15 letter or more decrease from baseline in best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity that is sustained for the participant's last 6 months of study participation. ETDRS visual acuity uses an eye chart with 5 letters per line. The scores range from 0 (no letters read correctly) to 100 (all letters read correctly).
Time Frame: Baseline through 48 months
Population: All randomized participants who took at least 1 dose of study drug and had post-baseline SMVL measurements.
Measure: Number; unit: percent of participants
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 146 | 138
percent of participants | 3.4 | 2.2
Statistical Analysis 1: Comparison: Placebo vs Ruboxistaurin; Test type: Superiority or Other; p = 0.724, Fisher Exact; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.15 to 2.67]

2. Secondary Outcome: Change From Baseline to Month 24 in Mean Retinal Thickness Within 500 Microns of the Center of the Macula
Description: Least Squares (LS) Mean values were controlled for treatment, pooled center, and baseline value.
Time Frame: Baseline, 24 months
Population: All randomized participants who took at least 1 dose of study drug and had both baseline and post-baseline retinal thickness measurements.
Measure: Least Squares Mean (Standard Error); unit: micrometer (µm)
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 148 | 149
micrometer (µm) | 12.8 (5.5) | 9.4 (5.3)
Statistical Analysis 1: Comparison: Placebo vs Ruboxistaurin; Test type: Superiority or Other; p = 0.616, Mixed models repeated measures; LS Mean difference = -3.3, 95% CI 2-sided [-16.5 to 9.8]

3. Secondary Outcome: Number of Eyes With Significant Center-Involved Macular Edema at Any Time From Baseline Through Month 24
Description: Significant center-involved macular edema is defined as an absolute retinal thickness at the center of the macula >2 standard deviations above the mean baseline value (where the mean and standard deviation are calculated at baseline from the randomized population of participants with retinal thickness values of ≤ 300 microns in depth).
Time Frame: Baseline through 24 months
Population: All randomized participants who took at least 1 dose of study drug and had post-baseline macular edema measurements.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 148 | 149
Number analyzed (Eyes) | 286 | 286
Eyes | 77 | 76
Statistical Analysis 1: Comparison: Placebo vs Ruboxistaurin; Test type: Superiority or Other; p = 0.971, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.68 to 1.44]

4. Secondary Outcome: Time to Focal Photocoagulation
Time Frame: Baseline through 48 months
Population: All randomized participants who took at least 1 dose of study drug and had post-baseline determination of focal photocoagulation treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 148 | 149
months | NA [NA to NA] — Median value was not calculable due to low number of participants requiring focal photocoagulation during the study. | NA [NA to NA] — Median value was not calculable due to low number of participants requiring focal photocoagulation during the study.

5. Secondary Outcome: Change From Baseline to Month 24 in Contrast Sensitivity
Description: Values are presented as changes in the number of letters read correctly on the Pelli-Robson contrast sensitivity chart which consists of 16 triplets (48 letters total) with letters of the same size but decreasing contrast. Least Squares (LS) Mean values were controlled for treatment, pooled center, and baseline value.
Time Frame: Baseline, 24 months
Population: All randomized participants who took at least 1 dose of study drug and had both baseline and post-baseline contrast sensitivity measurements.
Measure: Least Squares Mean (Standard Error); unit: letters read correctly
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 148 | 149
letters read correctly | -1.1 (0.4) | -0.6 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Ruboxistaurin; Test type: Superiority or Other; p = 0.344, Mixed models repeated measures; LS Mean difference = 0.5, 95% CI 2-sided [-0.6 to 1.6]

6. Secondary Outcome: Change From Baseline to Month 24 in Retinal Thickness at the Center of the Macula
Time Frame: Baseline, up to 24 months
Population: All randomized participants who took at least 1 dose of study drug and had both baseline and post-baseline retinal thickness measurements, last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: micrometer (µm)
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 148 | 149
micrometer (µm) | 10.5 (65.4) | 13.1 (74.9)
Statistical Analysis 1: Comparison: Placebo vs Ruboxistaurin; Test type: Superiority or Other; p = 0.663, ANCOVA

7. Secondary Outcome: Number of Participants Requiring Focal Photocoagulation at Any Time From Baseline Through Month 24
Time Frame: Baseline through 24 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 148 | 149
participants | 35 | 26
Statistical Analysis 1: Comparison: Placebo vs Ruboxistaurin; Test type: Superiority or Other; p = 0.203, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.37 to 1.23]

8. Secondary Outcome: Number of Participants Not Requiring Focal Photocoagulation at Any Time From Baseline Through Month 24
Time Frame: Baseline through 24 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 148 | 149
participants | 113 | 123

9. Secondary Outcome: Number of Participants Requiring Repeat Focal Photocoagulation at Any Time From Baseline Though Month 24
Description: Repeat focal photocoagulation is defined as 2 or more focal photocoagulation treatments needed during the study.
Time Frame: Baseline through 24 months
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | Ruboxistaurin
Number analyzed (Participants) | 148 | 149
participants | 11 | 12
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.749, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.46 to 2.92]

ADVERSE EVENTS:
Arm/Group | Placebo | Ruboxistaurin
Serious Adverse Events (participants affected / at risk) | 31/153 | 36/149
Other Adverse Events (participants affected / at risk) | 112/153 | 118/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | Ruboxistaurin (N=149)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (2)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Omphalitis (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 5 (5)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (4)
Wound infection (Infections and infestations) | 2 (3) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hiv test positive (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (6)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | Ruboxistaurin (N=149)
Cataract (Eye disorders) | 6 (7) | 5 (10)
Lacrimation increased (Eye disorders) | 5 (6) | 0 (0)
Vision blurred (Eye disorders) | 5 (6) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 13 (15)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (6) | 6 (7)
Pyrexia (General disorders) | 7 (10) | 6 (9)
Bronchitis (Infections and infestations) | 5 (5) | 4 (4)
Influenza (Infections and infestations) | 14 (20) | 7 (7)
Localised infection (Infections and infestations) | 7 (8) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (10) | 13 (20)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 3 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11 (11) | 4 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4)
Dizziness (Nervous system disorders) | 5 (7) | 3 (3)
Headache (Nervous system disorders) | 13 (17) | 14 (17)
Neuropathy peripheral (Nervous system disorders) | 5 (5) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Hypertension (Vascular disorders) | 14 (15) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days